CLINICAL TRIAL: NCT07244653
Title: Effect of Hologram Application During Burn Dressing on Pain, Anxiety, Fear, Patient Satisfaction, and Physiological Parameters: A Randomized Controlled Trial
Brief Title: Hologram Burn Dressing on Pain, Anxiety, Fear, Patient Satisfaction, and Physiological Parameters
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gamze BULUT (Other)
Collaborators: Ataturk University (Other)
Responsible Party: Sponsor-Investigator, Gamze BULUT, Research Assistant, Department of Surgical Nursing, Ataturk University
Organization: Ataturk University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: TAUNI-BURNHOLO-2025-RCT01
Record Dates: First submitted 2025-11-14; First posted 2025-11-24 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Anxiety; Burn Pain; Burn Patients; Fear
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control: Standard nursing care (No Intervention): Refers to routine, evidence-based, and protocol-driven nursing procedures performed during burn dressing without any additional non-pharmacological interventions. This includes wound cleaning, dressing application, patient monitoring, pharmacological pain management as prescribed, and therapeutic communication supported by institutional burn care guidelines.
- Intervention (Experimental): Hologram Application During Burn Dressing
  Interventions: Other: Showing videos with holograms

INTERVENTIONS:
Other: Showing videos with holograms — The intervention in this study is the use of a three-dimensional hologram video as a distraction method during burn dressing procedures.
  Unlike conventional video or virtual reality (VR) applications, the hologram projects interactive 3D images into real space without requiring headsets or wearable devices. Patients can visually perceive the holographic content directly in front of them, allowing natural interaction and immersion. This feature provides a stronger distraction effect by engaging the patient's attention with vivid and dynamic images during the painful procedure.
  Thus, the hologram differs from standard video watching by offering an immersive, spatial, and realistic experience that does not restrict movement or require equipment contact with the burned area.
  Arms: Intervention

SUMMARY:
Burn injuries are a significant global health problem, leading to serious physical, psychological, and social challenges for affected individuals. The literature emphasizes that dressing changes are among the most painful and anxiety-provoking procedures, negatively impacting treatment adherence and patient well-being. Although pharmacological methods are used to alleviate pain and anxiety, they are often insufficient due to potential side effects and addiction risks.

In recent years, advancements in digital technologies-particularly virtual reality (VR), augmented reality (AR), and hologram applications-have offered promising distraction-based approaches. Hologram technology, through three-dimensional and interactive visuals, can divert the patient's attention from traumatic stimuli, thereby reducing pain, anxiety, and fear in an innovative way. However, there is limited scientific evidence regarding the use of hologram applications during burn dressing changes.

This study aims to examine the effects of hologram applications on pain, anxiety, fear, patient satisfaction, and physiological parameters during burn dressing procedures. The research will be conducted at Erzurum City Hospital Burn Center, with a total of 70 patients assigned to experimental and control groups using simple randomization. Data collection tools will include the Visual Analogue Scale (VAS), the State-Trait Anxiety Inventory (STAI), the Burn Specific Pain Anxiety Scale, satisfaction and fear VAS assessments, and physiological parameter recording forms. The study will be carried out between November 2025 and May 2026. The results are expected to provide evidence-based insights into the feasibility and effectiveness of hologram technology as a non-pharmacological, innovative intervention in burn care.

DETAILED DESCRIPTION:
Burn injuries represent a major global health concern, resulting in substantial physical, psychological, and social burden for individuals. Among the therapeutic procedures applied in burn care, dressing changes are consistently reported as one of the most painful and anxiety-inducing interventions. These procedures may negatively influence treatment adherence, prolong recovery, and reduce the overall quality of life for patients. While pharmacological agents are commonly administered to reduce pain and anxiety during burn dressing, they may fail to provide adequate relief and can be associated with undesirable side effects and drug dependency risks. Therefore, there is a growing emphasis on complementary, non-pharmacological strategies that can enhance patient comfort and procedural tolerance.

With rapid advances in digital health technologies, immersive visual distraction methods such as virtual reality (VR), augmented reality (AR), and hologram-based systems have emerged as novel interventions in clinical settings. Hologram technology, which presents interactive three-dimensional images, may effectively shift the patient's focus away from traumatic procedures and reduce negative emotional responses. This innovative technique has the potential to minimize pain, anxiety, and fear by engaging cognitive and sensory pathways associated with distraction. Despite its promising nature, current scientific evidence regarding hologram applications during burn dressing changes remains limited, and there is a lack of controlled clinical trials evaluating its efficacy.

This randomized controlled study aims to investigate the effects of hologram application during burn dressing procedures on pain, anxiety, fear, patient satisfaction, and physiological responses. The study will be conducted with 70 patients receiving treatment at the Burn Center of Erzurum City Hospital. Participants will be randomly assigned to the experimental group, in which hologram technology will be applied during dressing changes, or to the control group receiving standard care. Data will be collected using validated tools including the Visual Analogue Scale (VAS) for pain and satisfaction, the Burn Specific Pain Anxiety Scale, the State-Trait Anxiety Inventory (STAI), fear assessment through VAS, and physiological monitoring forms for parameters such as heart rate, respiratory rate, and blood pressure. The research will be carried out between November 2025 and May 2026.

The findings of this study are expected to contribute high-quality evidence on the impact of hologram-based distraction as a non-pharmacological intervention in burn care. Results may support the integration of hologram technology into clinical practice to promote patient comfort, reduce emotional distress, and enhance overall treatment experience during burn dressing procedures.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 65,
* Able to read, write, and speak Turkish,
* Not participating in any other clinical trials at the same time,
* Patients who were decided to be admitted to a burn unit,
* No infected cases,
* Patients who did not undergo minor and/or major surgical procedures that could affect the wound healing process,
* No chronic illness other than burns,
* No cognitive, sensory, or other problems that would prevent verbal communication and understanding the information given,
* Second-degree burn with a total body surface area (TBSA) of less than 20%; Patients were included in the study if their burn rate was below 15% (20% in Grade 2 patients; sedation was required in Grade 3 patients with burn rates above 15%),
* 2nd and 3rd degree burns in the granulation stage (2nd and 3rd degree burns requiring granulation treatment and experiencing high pain),
* No burns on the head, ears, or face,
* Daily dressing changes with a frequency of 1-15 dressing changes,
* No complaints that would prevent participation in the study, such as respiratory problems,
* No vision or hearing problems.

Exclusion Criteria:

* Those with a pain intensity between 8 and 10 points (sedation is required when the pain intensity is 8 or higher),
* Those under the influence of various non-pharmacological treatment methods that may affect pain,
* Patients requiring advanced surgical procedures such as fasciotomy, escharotomy, or amputation,
* Patients receiving sedation during the dressing,
* Patients interrupting the hologram video during the dressing,
* First-degree burns,
* Those with neurological, psychological, or psychiatric illnesses,
* Patients receiving sedation during the dressing,
* Patients interrupting the hologram video during the dressing

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2026-06-20 (Estimated); Study Completion 2026-07-20 (Estimated)

PRIMARY OUTCOMES:
Pain intensity during burn dressing procedure | Immediately after the first and second dressing procedures (approximately 15-30 minutes each).
  Pain intensity will be assessed using the Visual Analogue Scale (VAS) ranging from 0 to 10, where **0 indicates "no pain" and 10 indicates "the worst possible pain." Higher scores indicate greater pain intensity.
State-Trait anxiety level | Immediately after the first and second dressing changes.
  State anxiety will be assessed using the State subscale of the State-Trait Anxiety Inventory (STAI-S). The scale ranges from 20 to 80 points, where higher scores indicate greater anxiety levels, and lower scores indicate reduced anxiety.
Burn-specific pain-related anxiety | Immediately after the first and second dressing procedures.
  Burn-specific pain-related anxiety will be assessed using the Burn Specific Pain Anxiety Scale (BSPAS). The scale ranges from 0 to 4 for each item, with a total score range of 0-64. Higher scores indicate greater levels of pain-related anxiety associated with burn procedures, while lower scores indicate reduced anxiety.
Fear level | Immediately after the first and second dressing procedures.
  Fear will be assessed using the Visual Analogue Scale (VAS) for Fear, ranging from 0 to 10, where **0 indicates "no fear" and 10 indicates "the highest possible fear." Higher scores indicate greater fear intensity.
Patient satisfaction | Immediately after the first and second dressing procedures.
  Patient satisfaction will be evaluated using the Visual Analogue Scale (VAS) for Satisfaction, ranging from 0 to 10, where **0 indicates "no satisfaction" and 10 indicates "maximum satisfaction." Higher scores indicate greater satisfaction with the dressing procedure.
Physiological parameter: Heart rate | Within each of the first and second dressing sessions (approximately 15-30 minutes).
  Heart rate will be measured using a standard patient monitor and recorded before, during, and immediately after each dressing procedure. Heart rate will be reported in beats per minute (bpm), where higher values indicate increased physiological stress, and lower values indicate reduced stress response.
Physiological parameter: Oxygen saturation | Within each of the first and second dressing sessions (approximately 15-30 minutes).
  Oxygen saturation will be measured using a standard patient monitor and reported as percentage (%) of oxygenated hemoglobin (SpO₂). Lower values may indicate higher physiological stress or discomfort, whereas higher values indicate better physiological stability.

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data (IPD) will not be shared due to patient privacy protection, ethical considerations, and institutional restrictions.